CLINICAL TRIAL: NCT02004691
Title: A Phase 2/3, Multicenter, Randomized, Double-blinded, Placebo-controlled, Repeat-dose Study to Evaluate the Efficacy, Safety, Pharmacodynamics, and Pharmacokinetics of Olipudase Alfa in Patients With Acid Sphingomyelinase Deficiency
Brief Title: Efficacy, Safety, Pharmacodynamic, and Pharmacokinetics Study of Olipudase Alfa in Patients With Acid Sphingomyelinase Deficiency
Acronym: ASCEND
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFI12712; U1111-1142-5963 (Registry Identifier: ICTRP); DFI12712 (Other: Sanofi Identifier); 2015-000371-26 (EudraCT Number)
Expanded Access: NCT04877132 (Approved for marketing)
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Results first posted 2022-05-24 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Sphingomyelin Lipidosis
MeSH Terms: conditions — Niemann-Pick Disease, Type A | interventions — Sodium Chloride; olipudase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (saline) administered intravenously once every 2 weeks during the 52 weeks of the primary analysis period for patients randomized to placebo.
  Interventions: Drug: placebo (saline)
- Olipudase alfa (Experimental): Olipudase alfa dose (3 mg/kg body weight) in saline administered intravenously once every 2 weeks during the 52 weeks of the primary analysis period for patients randomized to olipudase alfa, and during the extension treatment period for all patients.
  Interventions: Drug: Olipudase alfa

INTERVENTIONS:
Drug: placebo (saline) — Pharmaceutical form: solution administered once every two weeks during the 52 weeks of the primary analysis period for participants randomized to placebo.
  Route of administration: intravenous infusion
  Arms: Placebo
Drug: Olipudase alfa — Pharmaceutical form: Powder for concentrate for solution for infusion administered once every two weeks during the 52 weeks of the primary analysis period for participants randomized to olipudase alfa, and during the extension treatment period for all participants.
  Route of administration: intravenous infusion
  Other Names: GZ402665, Xenpozyme™
  Arms: Olipudase alfa

SUMMARY:
Primary Objective:

The primary objective of this phase 2/3 study was to evaluate the efficacy of olipudase alfa (recombinant human acid sphingomyelinase) administered intravenously once every 2 weeks for 52 weeks in adult participants with acid sphingomyelinase deficiency (ASMD) by assessing changes in: 1) spleen volume as measured by abdominal magnetic resonance imaging (MRI) (and, for the United States [US] only, in association with participant perception related to spleen volume as measured by splenomegaly-related score [SRS]); and 2) infiltrative lung disease as measured by the pulmonary function test, diffusing capacity of the lung for carbon monoxide (DLCO).

Secondary Objectives:

* To confirm the safety of olipudase alfa administered intravenously once every 2 weeks for 52 weeks.
* To characterize the effect of olipudase alfa on the participant perception related to spleen volume as measured by the SRS after 52 weeks of study drug administration. (For the US, the effect of olipudase alfa on the SRS is part of the primary objective).
* To characterize the effect of olipudase alfa after 52 weeks of study drug administration on the following outcome measures assessed sequentially:

  * The effect of olipudase alfa on liver volume;
  * The effect of olipudase alfa on platelet count;
  * The effect of olipudase alfa on fatigue;
  * The effect of olipudase alfa on pain;
  * The effect of olipudase alfa on dyspnea.

DETAILED DESCRIPTION:
The planned total duration per participant was for at least 3 years and up to 5 years and 3 months. This included up to approximately two month of screening, 52 weeks of primary analysis period, up to 4 years and 3 months of extension treatment period, an end-of- study visit within 2 weeks of the last treatment, and a safety follow-up 30 to 37 days after the last treatment.

ELIGIBILITY:
Inclusion criteria :

* The participant was willing and able to provide signed written informed consent.
* The participant was male or female aged 18 years or older.
* The participant had documented deficiency of acid sphingomyelinase as measured in peripheral leukocytes, cultured fibroblasts, or lymphocytes; and a clinical diagnosis consistent with Niemann-Pick disease type B (NPD B).
* The participant had diffuse capacity of the lung for carbon monoxide less than or equal to (<=)70% of the predicted normal value.
* The participant had a spleen volume greater than or equal to (>=)6 multiples of normal (MN) measured by MRI; participant who have had partial splenectomy was allowed if the procedure was performed >=1 year before screening/baseline and the residual spleen volume was >=6 MN.
* The participant had an SRS >=5.
* Female participants of childbearing potential must have had a negative serum pregnancy test for beta-human chorionic gonadotropin (β-HCG).
* Female participants of childbearing potential and male participants were willing to practice true abstinence in line with their preferred and usual lifestyle, or use 2 acceptable effective methods of contraception for up to 15 days following their last dose of study drug.

Exclusion criteria:

* The participant had received an investigational drug within 30 days before study enrollment.
* The participant had a medical condition, including significant intercurrent illness; significant cardiac disease (e.g., clinically significant arrhythmia, moderate or severe pulmonary hypertension or clinically significant valve dysfunction, or less than or equal to (<=)40% left ventricular ejection fraction by echocardiogram); active hepatitis B or hepatitis C, or infection with human immunodeficiency virus (HIV); malignancy diagnosed within the past 5 years (other than non-melanoma skin cancer), or any other serious medical condition that might have precluded participation in the study.
* The participant had a platelet count less than (<)60,000/microliters based on the average of 2 samples.
* The participant had an international normalized ratio (INR) greater than (>)1.5.
* The participant had alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >250 IU/L or total bilirubin >1.5 mg/dL (except for participant with Gilbert's syndrome).
* The participant had a major organ transplant (eg, bone marrow or liver).
* The participant was scheduled during the study for in-patient hospitalization including elective surgery and excluding the liver biopsies required per protocol.
* The participant, in the opinion of the investigator, was unable to adhere to the requirements of the study.
* The participant was unwilling or unable to abstain from the use of alcohol for 1 day before and 3 days after each study drug infusion. Testing for blood alcohol levels was not required.
* The participant was unwilling or unable to avoid 10 days before and 3 days after the protocol scheduled liver biopsies the use of medications or herbal supplements that were potentially hepatotoxic (e.g., 3-hydroxy-3-methyl glutaryl coenzyme A reductase inhibitors, erythromycin, valproic acid, anti-depressants, kava, echinacea) and/or might have caused or prolonged bleeding (e.g., anti-coagulants, ibuprofen, aspirin, garlic supplements, ginkgo, ginseng).
* The participant required medications that might have decreased olipudase alfa activity (e.g., fluoxetine, chlorpromazine, tricyclic antidepressants [e.g., imipramine, or desipramine]).
* The participant required use of invasive ventilatory support.
* The participant required use of noninvasive ventilator support while awake for longer than 12 hours daily.
* The participant was breast-feeding.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (24):
- United States (3):
  - UCSF Medical Center Site Number : 840005, San Francisco, California
  - Emory University Site Number : 840003, Decatur, Georgia
  - Montefiore Medical Center Site Number : 840006, The Bronx, New York
- Investigational Site Number : 032001, Córdoba, Argentina
- Investigational Site Number : 036001, Westmead, New South Wales, Australia
- Investigational Site Number : 056001, Leuven, Belgium
- Hospital De Clinicas De Porto Alegre Site Number : 076001, Porto Alegre, Rio Grande do Sul, Brazil
- Investigational Site Number : 100001, Sofia, Bulgaria
- Investigational Site Number : 152001, Santiago, Reg Metropolitana de Santiago, Chile
- Investigational Site Number : 250001, Paris, France
- Investigational Site Number : 276001, Mainz, Germany
- Italy (2):
  - Investigational Site Number : 380002, Napoli
  - Investigational Site Number : 380001, Udine
- Investigational Site Number : 392001, Fukushima, Fukushima, Japan
- Investigational Site Number : 528001, Amsterdam, Netherlands
- Investigational Site Number : 620002, Porto, Portugal
- Investigational Site Number : 724001, Madrid, Spain
- Investigational Site Number : 788001, Tunis, Tunisia
- Turkey (Türkiye) (4):
  - Investigational Site Number : 792002, Ankara
  - Investigational Site Number : 792004, Istanbul
  - Investigational Site Number : 792003, Istanbul
  - Investigational Site Number : 792001, Izmir
- United Kingdom (2):
  - Investigational Site Number : 826001, London, London, City of
  - Investigational Site Number : 826002, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.

REFERENCES:
- [Derived] Wasserstein MP, Lachmann R, Hollak C, Barbato A, Gallagher RC, Giugliani R, Guelbert NB, Hennermann JB, Ikezoe T, Lidove O, Mabe P, Mengel E, Scarpa M, Senates E, Tchan M, Villarrubia J, Thurberg BL, Yarramaneni A, Armstrong NM, Kim Y, Kumar M. Continued improvement in disease manifestations of acid sphingomyelinase deficiency for adults with up to 2 years of olipudase alfa treatment: open-label extension of the ASCEND trial. Orphanet J Rare Dis. 2023 Dec 2;18(1):378. doi: 10.1186/s13023-023-02983-0. PMID 38042851

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 23 active centers in 17 countries. A total of 62 participants were screened between 18 December 2015 and 22 October 2018, out of which 36 participants were randomized.
Pre-assignment Details: A total of 36 participants were randomized in a 1:1 ratio to receive either placebo or olipudase alfa in the primary analysis period (PAP) for 52 weeks. After completing PAP, participants entered an extension treatment period (ETP) where all participants received olipudase alfa up to Year 5.
Groups:
- Placebo: Participants received intravenous (IV) infusion of placebo (matched to olipudase alfa) once every 2 weeks up to Week 52. Participants who completed PAP entered in ETP and crossed over to olipudase alfa with a target maintenance dose of 3 mg/kg after dose escalation which was administered IV once every 2 weeks up to Year 5.
- Olipudase Alfa: Participants received IV infusion of olipudase alfa once every 2 weeks up to Week 52. Each participant underwent a dose escalation according to the following paradigm: 0.1, 0.3, 0.3, 0.6, 0.6, 1.0, 2.0, 3.0, 3.0 mg/kg. Three (3) mg/kg was the target maintenance dose, which was maintained for the remaining duration of 52 weeks of PAP. Participants who completed PAP entered in ETP and continued the same treatment in ETP up to Year 5.
Period: PAP: Up to 52 Weeks
Arm/Group | Placebo | Olipudase Alfa
Started | 18 | 18
Completed | 17 | 18
Not Completed | 1 | 0
Not completed — Poor compliance | 1 | 0
Period: ETP: From Week 52 up to 5 Years
Arm/Group | Placebo | Olipudase Alfa
Started | 17 | 18
Completed | 13 | 16
Not Completed | 4 | 2
Not completed — Related to Coronavirus Disease (COVID-19) | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Adverse Event not Related to COVID-19 | 1 | 0
Not completed — Not Related to COVID-19 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on modified intent-to-treat (mITT) population which included all randomized participants who had received at least 1 infusion (partial or total) and were analyzed according to the treatment arm allocated by randomization.
Groups:
- Placebo: Participants received IV infusion of placebo (matched to olipudase alfa) once every 2 weeks up to Week 52. Participants who completed PAP entered in ETP and crossed over to olipudase alfa with a target maintenance dose of 3 mg/kg after dose escalation which was administered IV once every 2 weeks up to Year 5.
Arm/Group | Placebo | Olipudase Alfa | Total Title
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.46 (17.06) | 36.17 (12.72) | 34.81 (14.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 5 | 9 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Black or African American | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Predicted (% Predicted) Hemoglobin (Hb) and Altitude-Adjusted Diffusing Capacity of the Lung for Carbon Monoxide (DLco) at Baseline
Description: Percent predicted Hb and Altitude-adjusted DLco was calculated as: 100*Adjusted DLco/Predicted DLco in unit of mL CO/min/mmHg where, adjusted DLco = Observed DLco (in mL CO/min/mmHg) times Hemoglobin-adjusted factor times Altitude-adjustment factor.
Time Frame: Baseline (Day 1)
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Deviation); unit: % Predicted DLco
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 18 | 18
% Predicted DLco | 48.45 (10.76) | 49.44 (10.99)

2. Primary Outcome: Percent Change From Baseline in Percent Predicted (% Predicted) Hemoglobin (Hb) and Altitude-Adjusted Diffusing Capacity of the Lung for Carbon Monoxide (DLco) at Week 52
Description: as for outcome 1
Time Frame: Baseline, Week 52
Population: Analysis was performed on mITT population. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 17 | 17
percent change | 2.961 (3.3832) | 21.968 (3.3362)
Statistical Analysis 1: Comparison: Placebo vs Olipudase Alfa; Test type: Superiority; p = 0.0004, Mixed model for repeated measures — Threshold for significance was 0.05; Least Squares Mean Difference = 19.008, 95% CI 2-sided [9.319 to 28.696], Standard Error of Mean 4.7576 — The 95% Confidence Interval (CI) and p-values were based on mixed model for repeated measures approach with Baseline Derived % Predicted DLco adjusted for Hb and pressure, age, treatment group, visit, and study visit by treatment group as covariates

3. Primary Outcome: Combination Spleen Endpoint: Component 1: Spleen Volume (in MN) at Baseline
Description: Spleen volume was assessed by abdominal magnetic resonance imaging (MRI) to quantitate the degree of splenomegaly in multiples of normal (MN).
Time Frame: Baseline (Day 1)
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Deviation); unit: multiples of normal (MN)
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 18 | 18
multiples of normal (MN) | 11.21 (3.84) | 11.69 (4.92)

4. Primary Outcome: Combination Spleen Endpoint: Component 1: Percent Change From Baseline in Spleen Volume (in MN) at Week 52
Description: Spleen volume was assessed by abdominal MRI to quantitate the degree of splenomegaly in MN.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 17 | 18
percent change | 0.481 (2.5002) | -39.446 (2.4294)
Statistical Analysis 1: Comparison: Placebo vs Olipudase Alfa; Test type: Superiority; p < .0001, Mixed model for repeated measures — Threshold for significance was 0.05; Least Squares Mean Difference = -39.927, 95% CI 2-sided [-47.051 to -32.803], Standard Error of Mean 3.4957 — The 95% CI and p-values were based on a mixed model for repeated measures approach with Baseline Spleen Volume (MN), Baseline age, treatment group, study visit, and study visit by treatment group interaction as covariates

5. Primary Outcome: Combination Spleen Endpoint (Primary for US Only): Component 2: Splenomegaly-Related Score (SRS) at Baseline
Description: The SRS rates 5 items: abdominal pain, abdominal discomfort, early satiety, dissatisfaction with abdominal body image, and difficulty to bend down using a numerical rating scale of 0 (absent) to 10 (worst imaginable). The total score of SRS ranges from 0 to 50, with higher scores (50) indicated worst imaginable rating. It was pre-specified as secondary endpoint for countries outside of US.
Time Frame: Baseline (Day 1)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 17 | 18
score on a scale | 28.05 (10.56) | 24.55 (11.13)

6. Primary Outcome: Combination Spleen Endpoint (Primary for US Only): Component 2: Change From Baseline in Splenomegaly-Related Score (SRS) at Week 52
Description: as for outcome 5
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 17 | 17
score on a scale | -9.281 (2.4165) | -7.664 (2.3481)
Statistical Analysis 1: Comparison: Placebo vs Olipudase Alfa; Test type: Superiority; p = 0.6364, Mixed model for repeated measures — Threshold for significance was 0.15; Least Squares Mean Difference = 1.618, 95% CI 2-sided [-5.302 to 8.538], Standard Error of Mean 3.3877 — The 95% CI and p-values are based on a mixed model for repeated measures approach with Baseline Splenomegaly Related Score, Baseline age, treatment group, study visit, and study visit by treatment group interaction as covariates

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) up to Week 52
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered with a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. TESAEs was defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. Reported AEs are treatment-emergent AEs that developed, worsened or became serious during the treatment period.
Time Frame: From the first infusion of investigational medicinal product (IMP) up to 52 weeks
Population: The safety population was a subset of the randomized population and included randomized participants who received at least 1 infusion (partial or total).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 18 | 18
Participants
  TEAEs | 18 | 18
  TESAEs | 4 | 3

8. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs) up to Week 52
Description: An AESI was defined as an AE (serious or nonserious) of scientific and medical concern specific to sponsor's product or program, for which ongoing monitoring and rapid communication by investigator to sponsor was appropriate. AESIs included any pregnancy, symptomatic overdose, dose-limiting toxicities (DLTs) as defined in protocol and infusion associated reactions (IARs). Protocol-defined IARs were AEs that occurred during the infusion or within up to 24 hours after the start of infusion and were considered as related or possibly related to the study treatment by the investigator or the sponsor. Events occurring greater than or equal to (>=) 24 hours after the start of an infusion might have been judged an IAR at the discretion of the investigator or sponsor. Algorithm-defined IARs were all AEs that started between the start of infusion and the end of infusion plus 24 hours, irrespective of the perceived relation with study treatment.
Time Frame: From the first infusion of IMP up to 52 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 18 | 18
Participants
  Pregnancy | 0 | 0
  Symptomatic Overdose | 0 | 0
  DLTs | 5 | 1
  Protocol-defined IARs | 5 | 8
  Algorithm-defined IARs | 13 | 15

9. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities (PCSA) in Liver Function Tests up to Week 52
Description: PCSA criteria: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST): >3 x upper limit of normal (ULN), >5 x ULN, >10 x ULN and >20 x ULN. Alkaline phosphatase (ALP) > 1.5 x ULN. Total bilirubin >1.5 x ULN and >2 x ULN. ALT and total bilirubin: ALT > 3 x ULN and total bilirubin > 2 x ULN. Baseline was defined as the last non-missing value prior to the first infusion of study treatment.
Time Frame: From Baseline (Day 1) up to 52 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 18 | 18
Participants
  ALT: >3 x ULN | 2 | 1
  ALT: >5 x ULN | 1 | 1
  ALT: >10 x ULN | 0 | 0
  ALT: >20 x ULN | 0 | 0
  AST: >3 x ULN | 2 | 2
  AST: >5 x ULN | 1 | 1
  AST: >10 x ULN | 0 | 0
  AST: >20 x ULN | 0 | 0
  ALP: >1.5 x ULN | 1 | 1
  Total Bilirubin: >1.5 x ULN | 4 | 4
  Total Bilirubin: >2 x ULN | 1 | 4
  ALT >3 x ULN and total bilirubin >2 x ULN | 0 | 1

10. Secondary Outcome: Number of Participants Who Developed Anti-Drug Antibodies (ADA) to Olipudase Alfa up to Week 52
Description: Number of participants with treatment-emergent ADA are presented. Baseline was defined as the last non-missing value prior to the first infusion of study treatment.
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 18 | 18
Participants | 1 | 4

11. Secondary Outcome: Percent Change From Baseline in Liver Volume (in MN) at Week 52
Description: Liver volume was assessed by abdominal MRI in MN.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 17 | 18
percent change | -1.468 (2.5409) | -28.064 (2.4899)
Statistical Analysis 1: Comparison: Placebo vs Olipudase Alfa; A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in an order the outcome measure were reported and continued when previous endpoint was statistically significant at two-sided 0.05; Test type: Superiority; p < .0001, Mixed model for repeated measures — Threshold for significance was 0.05; Least Squares Mean Difference = -26.596, 95% CI 2-sided [-33.911 to -19.281], Standard Error of Mean 3.5862 — The 95% CI and p-values are based on a mixed model for repeated measures approach with Baseline Liver Volume (MN), Baseline age, treatment group, study visit, and study visit by treatment group interaction as covariates

12. Secondary Outcome: Percent Change From Baseline in Platelet Counts at Week 52
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 16 | 18
percent change | 2.490 (4.1923) | 16.822 (3.9596)
Statistical Analysis 1: Comparison: Placebo vs Olipudase Alfa; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0185, Mixed model for repeated measures — Threshold for significance was 0.05; Least Squares Mean Difference = 14.332, 95% CI 2-sided [2.564 to 26.099], Standard Error of Mean 5.7822 — The 95% CI and p-values are based on a mixed model for repeated measures approach with Baseline Platelets, Baseline age, treatment group, study visit, and study visit by treatment group interaction as covariates

13. Secondary Outcome: Change From Baseline in Fatigue Severity as Measured by Brief Fatigue Inventory (BFI)-Item 3 Scale Score at Week 52
Description: The BFI is a 9-item, validated, self-administered questionnaire that was originally developed to assess fatigue severity. The 9-items were measured on a 0-10 scale, with 0 being 'does not interfere' and 10 being 'completely interferes.' BFI - Item 3 asks participants to "Please rate your fatigue (weariness, tiredness) by circling the one number that best describes your worst level of fatigue during the past 24 hours. Numerical rating scale ranges from 0 (no fatigue) to 10 (worst imaginable fatigue). Higher global scores were associated with more severe fatigue.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 17 | 17
score on a scale | -1.806 (0.5272) | -1.862 (0.5129)
Statistical Analysis 1: Comparison: Placebo vs Olipudase Alfa; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.9400, Mixed model for repeated measures — Threshold for significance was 0.05; Least Squares Mean Difference = -0.056, 95% CI 2-sided [-1.566 to 1.454], Standard Error of Mean 0.7384 — The 95% CI and p-values are based on a mixed model for repeated measures approach with Baseline BFI item 3 (Worst Fatigue), Baseline age, treatment group, study visit, and study visit by treatment group interaction as covariates

14. Secondary Outcome: Change From Baseline in Pain Severity as Measured by Brief Pain Inventory-Short Form (BPI-SF)-Item 3 Scale Score at Week 52
Description: The BPI-SF is a validated, self-administered questionnaire designed to measure a participant's perceived level of pain. The BPI-SF consisted of 15 items that use a numeric rating scale to assess pain severity and pain interference in the past 24 hours and the past week. For BPI-SF Item 3 asks participants to "Please rate your pain by marking the box beside the number that best describes your pain at its worst in the past 24 hours." The numeric rating scale ranged from 0 (no pain) to 10 (worst imaginable pain), where higher scores indicate greater intensity of pain.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 17 | 17
score on a scale | -2.293 (0.5899) | -1.404 (0.5742)

15. Secondary Outcome: Change From Baseline in Dyspnea Severity as Measured by Functional Assessment of Chronic Illness Therapy (FACIT) Dyspnea Scale at Week 52
Description: FACIT-Dyspnea is a 20 Item assessment that is split into two 10-item sections. The first 10-item section asks participants about the severity of their shortness of breath during various activities. The second 10-item section asks participants to rate the difficulty due to shortness of breath associated with the same activities that were referenced in the first section. For the dyspnea severity items, score range from 0=no shortness of breath; 1=mildly short of breath; 2=moderately short of breath; 3=severely short of breath. For the functional limitation items, score range from no difficult = 0, A little difficult = 1, some difficult = 2, and much difficulty =3. A raw score was calculated as: sum of individual item scores * 10/number of items answered. Raw scores were then converted to scale scores using the table included in the FACIT Dyspnea Scale Short Form Scoring Guideline. FACIT dyspnea scale score ranged between 27.7 to 75.9. Higher score represented high levels of dyspnea.
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Olipudase Alfa
Number analyzed (Participants) | 11 | 16
score on a scale | -6.769 (1.9132) | -5.862 (1.6918)

ADVERSE EVENTS:
Time Frame: For PAP: From the first infusion of IMP up to 52 weeks. For ETP: From Week 52 up to 5 years
Description: Analysis was performed on safety population. MedDRA version 23.1 was used for PAP; whereas MedDRA version 26.0 was used for ETP data. Any non-serious AE with a preferred term in >= 2 % participants and number of participants >= 2 in the Olipudase Alfa group and the percentage of participants with the specific TEAE in the Olipudase Alfa group is greater than placebo group.
Groups:
- PAP: Placebo: Subjects received IV infusion of placebo (matched to olipudase alfa) once every 2 weeks up to Week 52.
- PAP: Olipudase Alfa: Subjects received IV infusion of olipudase alfa once every 2 weeks up to Week 52. Each subject underwent a dose escalation according to the following paradigm: 0.1, 0.3, 0.3, 0.6, 0.6, 1.0, 2.0, 3.0,3.0 mg/kg. Three (3) mg/kg was the target maintenance dose, which was maintained for the remaining duration of 52 weeks of PAP.
- ETP: Placebo/Olipudase Alfa: Subjects who completed PAP entered in ETP and crossed over to olipudase alfa with a target maintenance dose of 3 mg/kg after dose escalation which was administered IV once every 2 weeks up to Year 5.
- ETP: Olipudase Alfa/Olipudase Alfa: Subjects who completed PAP entered in ETP and continued the same treatment in ETP up to Year 5.
Arm/Group | PAP: Placebo | PAP: Olipudase Alfa | ETP: Placebo/Olipudase Alfa | ETP: Olipudase Alfa/Olipudase Alfa
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 4/18 | 3/18 | 6/17 | 5/18
Other Adverse Events (participants affected / at risk) | 13/18 | 17/18 | 9/17 | 12/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAP: Placebo (N=18) | PAP: Olipudase Alfa (N=18) | ETP: Placebo/Olipudase Alfa (N=17) | ETP: Olipudase Alfa/Olipudase Alfa (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic Haemorrhage (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastritis Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aortic Dilatation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis Superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAP: Placebo (N=18) | PAP: Olipudase Alfa (N=18) | ETP: Placebo/Olipudase Alfa (N=17) | ETP: Olipudase Alfa/Olipudase Alfa (N=18)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 7 (8) | 8 (9)
Nasopharyngitis (Infections and infestations) | 6 (8) | 8 (18) | 5 (10) | 7 (22)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (6) | 6 (8) | 3 (7) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (10) | 3 (5) | 1 (2)
Headache (Nervous system disorders) | 8 (32) | 12 (64) | 4 (48) | 5 (53)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (5) | 1 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT02004691/Prot_002.pdf
  • Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT02004691/SAP_001.pdf